CLINICAL TRIAL: NCT01014936
Title: A Phase I Open-label, Non-randomized, Dose-escalation First-in-man Trial to Investigate the c-Met Kinase Inhibitor MSC2156119J Under Three Different Regimens in Subjects With Advanced Solid Tumors
Brief Title: First-in-Man, Dose-escalation Trial of C-met Kinase Inhibitor MSC2156119J in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200095_001; 2013-003767-63 (EudraCT Number)
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Patients With Solid Tumors, Either Refractory to Standard Therapy or for Which no Effective Standard Therapy is Available
Keywords: Phase 1; advanced solid tumors; refractory to standard therapy
MeSH Terms: interventions — EMD1214063; tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MSC2156119J Regimen 1 (Experimental): Subjects will be administered with micronized or non-micronized MSC2156119J in dose ranging from 30 mg to 400 mg (capsule formulation) once daily for 14 days, followed by 7 days with no treatment (21-day cycle) in Regimen 1.
  Interventions: Drug: MSC2156119J
- MSC2156119J Regimen 2 (Experimental): Subjects will be administered with micronized or non-micronized MSC2156119J in dose ranging from 60 mg to 315 mg (capsule formulation) once daily 3 times per week for 3 weeks (21-day cycle) in Regimen 2.
  Interventions: Drug: MSC2156119J
- MSC2156119J Regimen 3 (Experimental): Subjects will be administered with micronized MSC2156119J in dose ranging from 300 mg to 1400 mg (capsule or tablet formulation) once daily for 21 days (21-day cycle) in Regimen 3.
  Interventions: Drug: MSC2156119J

INTERVENTIONS:
Drug: MSC2156119J
  Other Names: EMD 1214063; Tepotinib

SUMMARY:
This is a an open-label, dose-escalation, first-in-man (FIM) study designed to explore MSC2156119J, in subjects with advanced solid tumors who have not responded to previous therapies or for whom no other therapies are available.

Subjects will be assigned one of the dosing regimens:

* Regimen 1: MSC2156119J once daily for 14 days, followed by 7 days with no treatment (21-day cycle)
* Regimen 2: MSC2156119J three times per week (e.g., Days 1, 3, and 5) for three weeks (21-day cycle)
* Regimen 3: MSC2156119J every day for three weeks (21-day cycle)

ELIGIBILITY:
Inclusion Criteria:

1. Subject should read and fully understand the requirements of the trial, be willing to comply with all trial visits and assessments, and be willing and able to give informed consent
2. Histologically or cytologically confirmed solid tumor, either refractory to standard therapy or for which no effective standard therapy is available
3. Measurable or evaluable disease, as defined by RECIST 1.0
4. Estimated life expectancy greater than (>) three months
5. Men or women aged greater than or equal to (>=) 18 years
6. Women of childbearing potential must have a negative blood pregnancy test at the Screening Visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are post-menopausal for at least 12 months, are surgically sterile, or are sexually inactive.
7. Subjects and their partners must be willing to avoid pregnancy during the trial and until three months after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator, such as a two-barrier method or one-barrier method with spermicide or intrauterine device. This requirement begins two weeks before receiving the first trial treatment and ends one month after receiving the last treatment.
8. ECOG performance status of 0 to 2
9. Adequate hematological function:

   * Hemoglobin >= 9.0 g/dL
   * Neutrophils > 1.5 x 109/L
   * Platelets >= 75 x 109/L
10. Adequate liver function:

    * Total bilirubin less than or equal to (<=) 1.5 x ULN (upper limit to normal)
    * AST/ ALT ≤ 2.5 x ULN

    For subjects with liver metastases:
    * Total bilirubin ≤ 1.5 x ULN
    * AST/ ALT ≤ 5 x ULN
11. Adequate renal function:

    * Serum creatinine < 1.5 x ULN, and/or
    * Calculated creatinine clearance > 60 mL/min
12. Resolution of all acute chemotherapy, radiotherapy or surgery-related AEs to Grade <= 2, except for alopecia
13. Recovery from any surgical intervention
14. Subjects enrolling after the MTD has been determined must present specific c Met alterations (mutation, overexpression, amplification

Exclusion Criteria:

1. Received chemotherapy, immunotherapy, hormonal therapy (except subjects with prostate cancer), biologic therapy, or any other investigational agent or anticancer therapy within 28 days (or five half-lives for non-cytotoxics, whichever is shorter), of Day 1 of trial treatment (six weeks for nitrosureas or mitomycin C)
2. Received extensive prior radiotherapy on more than 30% of bone marrow
3. Symptomatic primary tumors or metastasis of brain and/or central nervous system, uncontrolled with antiepileptics and requiring high doses of steroids
4. Known HIV positivity, active hepatitis C, or active hepatitis B
5. Medical history of liver fibrosis/ cirrhosis
6. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
7. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product
8. Medical history of surgery within six weeks prior to enrollment
9. Impaired cardiac function (left ventricular ejection fraction < 45% defined by echocardiograph, serious arrhythmia, unstable angina pectoris, congestive heart failure NYHA III and IV, myocardial infarction within the last 12 months prior to trial entry; signs of pericardial effusion)
10. Hypertension uncontrolled by standard therapies (not stabilized to 150/90 mm Hg)
11. Peripheral neuropathy Grade >= 2
12. Medical history of any other significant medical disease, major surgery, or psychiatric condition that might impair the subject's well being or preclude full participation in the trial
13. Women who are pregnant or nursing
14. Known drug abuse or alcohol abuse
15. Participation in another clinical trial within the past 28 days
16. Requires concurrent treatment with a non-permitted drug
17. Known hypersensitivity to any of the trial treatment ingredients
18. Legal incapacity or limited legal capacity
19. Any other reason that, in the opinion of the principal investigator, precludes the subject from participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Falchook GS, Kurzrock R, Amin HM, Xiong W, Fu S, Piha-Paul SA, Janku F, Eskandari G, Catenacci DV, Klevesath M, Bruns R, Stammberger U, Johne A, Bladt F, Friese-Hamim M, Girard P, El Bawab S, Hong DS. First-in-Man Phase I Trial of the Selective MET Inhibitor Tepotinib in Patients with Advanced Solid Tumors. Clin Cancer Res. 2020 Mar 15;26(6):1237-1246. doi: 10.1158/1078-0432.CCR-19-2860. Epub 2019 Dec 10. PMID 31822497
- [Derived] Xiong W, Hietala SF, Nyberg J, Papasouliotis O, Johne A, Berghoff K, Goteti K, Dong J, Girard P, Venkatakrishnan K, Strotmann R. Exposure-response analyses for the MET inhibitor tepotinib including patients in the pivotal VISION trial: support for dosage recommendations. Cancer Chemother Pharmacol. 2022 Jul;90(1):53-69. doi: 10.1007/s00280-022-04441-3. Epub 2022 Jun 30. PMID 35771259
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR200095_001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First/last subject (informed consent): November 2009/December 2014. Last subject completed: October 2015. Clinical data cut-off: February 2016
Groups:
- MSC2156119J Regimen 1: Subjects were administered with micronized or non-micronized MSC2156119J in dose ranging from 30 mg to 400 mg (capsule formulation) once daily for 14 days, followed by 7 days with no treatment (21-day cycle) in Regimen 1.
- MSC2156119J Regimen 2: Subjects were administered with micronized or non-micronized MSC2156119J in dose ranging from 60 mg to 315 mg (capsule formulation) once daily 3 times per week for 3 weeks (21-day cycle) in Regimen 2.
- MSC2156119J Regimen 3: Subjects were administered with micronized MSC2156119J in dose ranging from 300 mg to 1400 mg (capsule or tablet formulation) once daily for 21 days (21-day cycle) in Regimen 3.
Period: Overall Study
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Started | 42 | 45 | 62
Completed | 42 | 45 | 62
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3 | Total
Number analyzed (Participants) | 42 | 45 | 62 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.97 (13.496) | 59.29 (14.656) | 56.49 (13.986) | 58.32 (14.050)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 25 | 66
  Male | 24 | 22 | 37 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Dose Limiting Toxicity (DLT)
Description: DLT was defined as one of the following adverse events (AEs) observed during Cycle1, regardless of MSC2156119J relationship, excluding AEs assessed by investigator exclusively related to subject's underlying disease or medical condition: Grade 4 neutropenia for >7 days; Grade >=3 febrile neutropenia for >1 day; Grade 4 thrombocytopenia/Grade 3 with bleeding; Grade >=3 nausea and emesis, despite optimal treatment; Grade >=3 non-hematological AE, except emesis and nausea with no adequate therapy and alopecia, Grade >= 3 liver AE with a recovery period of >7 days or to Grade <=1 for subjects without liver metastases or to <=2 for subjects with liver metastases; Grade >=3 lipase and/or amylase rise with pancreatitis confirmation, either based on clinical or radiological signs. Any AE not otherwise defined as a DLT that, due to prolonged recovery to Grade <=1 or baseline status, leads to delay of above 21 days in planned administration of study drug.
Time Frame: Day 1, 3, 8, 14, 17 of Cycle 1 (for Regimen 1 and 3); Day 1, 3, 8, 15, 19 of Cycle 1 (for Regimen 2)
Population: DLT analysis set comprised of subjects who had either completed Cycle 1 or had stopped treatment because of a DLT during Cycle 1.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 42 | 42 | 21
subjects | 1 | 3 | 2

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: MTD was defined as the dose level at which 2 out of 3 subjects or 2 out of 6 subjects experienced a DLT. The primary endpoint was to determine MTD of MSC2156119J for each of the 3 treatment regimens in subjects with advanced solid tumors. However, during the course of the trial it was established that the MTD could not be determined and instead, RP2D was to be determined.
Time Frame: Cycle 1 (Day 1 to Day 21)
Population: as for outcome 1
Measure: Number; unit: milligram
Groups:
- MSC2156119J Combined: All subjects who were administered with micronized or non-micronized MSC2156119J (capsule or tablet formulation) in any of the three regimens.
Arm/Group | MSC2156119J Combined
Number analyzed (Participants) | 105
milligram | 500

3. Primary Outcome: Number of Subjects With Treatment-Related Adverse Events
Description: Related AE was defined as any untoward medical occurrence which was considered to have a relationship with the study drug (suspected to be reasonably related to the study drug or AE was medically (pharmacologically/clinically) attributed to the study drug as per Investigator's assessment.
Time Frame: Baseline up to 158.01 weeks
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 42 | 45 | 62
subjects | 14 | 23 | 39

4. Secondary Outcome: Number of Subjects With Treatment-Emergent AEs (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation or TEAEs Leading to Death
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 33 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 158.01 weeks
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 42 | 45 | 62
subjects
  TEAEs | 41 | 45 | 59
  Serious TEAEs | 14 | 17 | 22
  TEAEs Leading to Discontinuation | 3 | 4 | 13
  TEAEs Leading To Death | 0 | 0 | 1

5. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Single Dose of MSC2156119J: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: Pharmacokinetic (PK) analysis set included all subjects who had received at least 1 dose of MSC2156119J and who had provided at least 1 concentration of MSC2156119J measurement after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- MSC2156119J 30 mg: Fed: Subjects were administered with micronized MSC2156119J 30 mg (capsule formulation) with food.
- MSC2156119J 60 mg: Fed: Subjects were administered with micronized MSC2156119J 60 mg (capsule formulation) with food.
- MSC2156119J 100 mg: Fed: Subjects were administered with micronized MSC2156119J 100 mg (capsule formulation) with food.
- MSC2156119J 145 mg: Fed: Subjects were administered with micronized MSC2156119J 145 mg (capsule formulation) with food.
- MSC2156119J 215 mg: Fed: Subjects were administered with micronized MSC2156119J 215 mg (capsule formulation) with food.
- MSC2156119J 300 mg: Fed: Subjects were administered with micronized MSC2156119J 300 mg (capsule formulation) with food.
- MSC2156119J 400 mg: Fed: Subjects were administered with micronized MSC2156119J 400 mg (capsule formulation) with food.
- MSC2156119J 30 mg: Fasted: Subjects were administered with non-micronized MSC2156119J 30 mg (capsule formulation) in the fasted state.
- MSC2156119J 60 mg: Fasted: Subjects were administered with non-micronized MSC2156119J 60 mg (capsule formulation) in the fasted state.
- MSC2156119J 115 mg: Fasted: Subjects were administered with non-micronized MSC2156119J 115 mg (capsule formulation) in the fasted state.
- MSC2156119J 115 mg: Fed: Subjects were administered with non-micronized MSC2156119J 115 mg (capsule formulation) with food.
- MSC2156119J 230 mg: Fasted: Subjects were administered with non-micronized MSC2156119J 230 mg (capsule formulation) in the fasted state.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 3
nanogram per milliliter (ng/mL) | 56.62 (20.4) | 70.65 (19.3) | 107.0 (29.6) | 147.0 (24.0) | 193.8 (55.3) | 306.4 (42.2) | 348.1 (18.6) | 3.445 (104.5) | 12.64 (44.5) | 13.72 (142.0) | 13.38 (74.1) | 29.03 (94.1)

6. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Single Dose of MSC2156119J: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: PK analysis set included all subjects who had received at least 1 dose of MSC2156119J and who had provided at least 1 concentration of MSC2156119J measurement after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC2156119J 130 mg: Fed: Subjects were administered with micronized MSC2156119J 130 mg (capsule formulation) with food.
- MSC2156119J 175 mg: Fed: Subjects were administered with micronized MSC2156119J 175 mg (capsule formulation) with food.
- MSC2156119J 315 mg: Fed: Subjects were administered with micronized MSC2156119J 315 mg (capsule formulation) with food.
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 3 | 4 | 6 | 7
ng/mL | 55.55 (53.6) | 115.5 (59.3) | 134.8 (22.3) | 142.4 (58.9) | 333.7 (78.5) | 5.926 (102.3) | 10.79 (67.1) | 22.24 (141.0) | 37.42 (64.4)

7. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Single Dose of MSC2156119J: Regimen 3
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC2156119J 500 mg: Fasted: Subjects were administered with micronized MSC2156119J 500 mg (capsule formulation) in the fasted state.
- MSC2156119J 500 mg: Fed: Subjects were administered with micronized MSC2156119J 500 mg (capsule formulation) with food.
- MSC2156119J 700 mg: Fed: Subjects were administered with micronized MSC2156119J 700 mg (capsule formulation) with food.
- MSC2156119J 1000 mg: Fed: Subjects were administered with micronized MSC2156119J 1000 mg (capsule formulation) with food.
- MSC2156119J 1200 mg: Fasted: Subjects were administered with micronized MSC2156119J 1200 mg (capsule formulation) in the fasted state.
- MSC2156119J 1400 mg: Fed: Subjects were administered with micronized MSC2156119J 1400 mg (capsule formulation) with food.
- MSC2156119J 500 mg: Fed (Tablet): Subjects were administered with micronized MSC2156119J 500 mg (tablet formulation) with food.
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 19 | 3 | 7 | 1 | 6 | 22
ng/mL | 246.5 (32.7) | 552.0 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 329.9 (72.4) | 433.5 (27.6) | 666.1 (46.0) | 761.0 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 863.4 (37.4) | 460.9 (58.7)

8. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Multiple Dose of MSC2156119J: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: PK analysis set included all subjects who had received at least 1 dose of MSC2156119J and who had provided at least 1 concentration of MSC2156119J measurement after the first dose. Here, "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3
ng/mL | 112.6 (26.1) | 204.6 (24.2) | 262.8 (10.2) | 379.3 (19.8) | 697.2 (49.8) | 810.9 (12.3) | 562.5 (45.0) | 28.54 (181.7) | 59.76 (110.0) | 48.33 (102.8) | 155.6 (249.6) | 210.1 (54.8)

9. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Multiple Dose of MSC2156119J: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3 | 3 | 3 | 6 | 6
ng/mL | 88.55 (53.0) | 181.4 (34.4) | 178.4 (67.6) | 300.5 (8.9) | 722.4 (32.2) | 8.458 (339.9) | 54.30 (48.5) | 52.30 (140.7) | 70.04 (68.5)

10. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) After Multiple Dose of MSC2156119J: Regimen 3
Description: Reporting group "MSC2156119J 1200 mg: Fasted" is not applicable for Multiple Dosing because only one subject was erroneously dosed with 1200 mg in fasted state as a single dose in Regimen 3. For multiple dose PK profile (Study Day 14), this subject was included in reporting group "MSC2156119J 1400 mg: Fed".
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 17 | 3 | 6 | 4 | 18
ng/mL | 741.6 (45.7) | 795.0 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 943.1 (34.6) | 1006 (39.4) | 1219 (59.2) | 1805 (31.2) | 1291 (48.1)

11. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Single Dose of MSC2156119J: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 3
hours | 8.000 [2.00 to 24.05] | 10.000 [8.00 to 24.00] | 10.000 [4.00 to 24.00] | 8.000 [8.00 to 10.00] | 8.000 [4.00 to 24.00] | 10.000 [4.10 to 24.00] | 8.000 [8.00 to 10.05] | 4.000 [4.00 to 10.00] | 8.000 [8.00 to 24.00] | 10.000 [4.00 to 24.00] | 24.000 [8.00 to 25.65] | 8.000 [4.00 to 24.00]

12. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Single Dose of MSC2156119J: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24, 48, 49.32 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 3 | 4 | 6 | 7
hours | 9.000 [4.00 to 24.20] | 8.000 [4.000 to 23.83] | 9.000 [4.03 to 24.33] | 8.000 [4.00 to 24.03] | 24.000 [7.97 to 24.03] | 10.000 [8.00 to 48.00] | 17.042 [8.00 to 48.00] | 33.083 [8.00 to 48.00] | 24.000 [8.00 to 49.32]

13. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Single Dose of MSC2156119J: Regimen 3
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Groups:
- MSC2156119J 500 mg Fed (Tablet): Subjects were administered with micronized MSC2156119J 500 mg (tablet formulation) with food.
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 19 | 3 | 7 | 1 | 6 | 22
hours | 8.000 [8.00 to 24.00] | 8.000 [8.00 to 8.00] | 10.000 [4.00 to 24.00] | 10.000 [4.00 to 24.00] | 10.000 [4.00 to 10.17] | 10.000 [10.00 to 10.00] | 24.000 [8.00 to 24.00] | 8.025 [4.00 to 24.10]

14. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Multiple Dose of MSC2156119J: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3
hours | 2.125 [0.00 to 4.25] | 8.000 [4.03 to 8.00] | 8.000 [4.00 to 24.00] | 4.000 [0.00 to 24.00] | 8.000 [4.00 to 8.00] | 8.000 [0.00 to 10.15] | 0.250 [0.00 to 10.00] | 4.000 [0.00 to 24.00] | 4.000 [0.00 to 8.00] | 6.000 [0.00 to 24.00] | 0.00 [0.00 to 0.00] | 4.000 [1.00 to 10.00]

15. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Multiple Dose of MSC2156119J: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Groups:
- MSC2156119J 130 mg Fed: Subjects were administered with micronized MSC2156119J 130 mg (capsule formulation) with food.
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3 | 3 | 3 | 6 | 6
hours | 10.000 [4.12 to 10.08] | 10.000 [2.00 to 24.13] | 8.000 [4.00 to 10.00] | 10.000 [8.00 to 10.00] | 8.000 [8.00 to 25.93] | 8.000 [8.00 to 24.00] | 8.067 [4.00 to 24.00] | 17.083 [8.00 to 24.08] | 10.000 [8.00 to 24.12]

16. Secondary Outcome: Time To Reach Maximum Plasma Concentration (Tmax) After Multiple Dose of MSC2156119J: Regimen 3
Description: as for outcome 10
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 17 | 3 | 6 | 4 | 18
hours | 10.000 [0.50 to 10.00] | 10.000 [10.00 to 10.00] | 8.000 [0.00 to 24.00] | 3.183 [0.25 to 8.00] | 8.833 [0.00 to 24.00] | 9.075 [2.83 to 24.00] | 8.000 [2.00 to 24.00]

17. Secondary Outcome: Apparent Terminal Half-life ( t1/2) After Single Dose Of MSC2156119J: Regimen 1
Description: Apparent Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of t1/2.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Apparent Terminal Half-life ( t1/2) After Single Dose Of MSC2156119J: Regimen 2
Description: as for outcome 17
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 17
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Apparent Terminal Half-life ( t1/2) After Single Dose Of MSC2156119J: Regimen 3
Description: as for outcome 17
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 17
Groups:
- MSC2156119J 300 mg Fed: Subjects were administered with micronized MSC2156119J 300 mg with food.
- MSC2156119J 500 mg Fasted: Subjects were administered with micronized MSC2156119J 500 mg in the fasted state.
- MSC2156119J 500 mg Fed: Subjects were administered with micronized MSC2156119J 500 mg with food.
- MSC2156119J 700 mg Fed: Subjects were administered with micronized MSC2156119J 700 mg with food.
- MSC2156119J 1000 mg Fed: Subjects were administered with micronized MSC2156119J 1000 mg with food.
- MSC2156119J 1200 mg Fasted: Subjects were administered with micronized MSC2156119J 1200 mg in the fasted state.
- MSC2156119J 1400 mg Fed: Subjects were administered with micronized MSC2156119J 1400 mg with food.
- MSC2156119J 500 mg Fed (Tablet): Subjects were administered with micronized MSC2156119J 500 mg (tablet) with food.
Arm/Group | MSC2156119J 300 mg Fed | MSC2156119J 500 mg Fasted | MSC2156119J 500 mg Fed | MSC2156119J 700 mg Fed | MSC2156119J 1000 mg Fed | MSC2156119J 1200 mg Fasted | MSC2156119J 1400 mg Fed | MSC2156119J 500 mg Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Apparent Terminal Half-life (t1/2) After Multiple Dose Of MSC2156119J: Regimen 1
Description: as for outcome 17
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 17
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Apparent Terminal Half-life (t1/2) After Multiple Dose Of MSC2156119J: Regimen 2
Description: as for outcome 17
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 17
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Apparent Terminal Half-life (t1/2) After Multiple Dose Of MSC2156119J: Regimen 3
Description: as for outcome 17
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 17
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve From Time Zero to Last Sampling Time (AUC0-t) After First Dose of MSC2156119J: Regimen 1
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- MSC2156119J 60 mg Fasted: Subjects were administered with non-micronized MSC2156119J 60 mg in the fasted state.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6
h*ng/mL | 849.4 (24.5) | 1283.0 (23.9) | 1433.5 (35.5) | 2532.7 (12.6) | 3105.5 (60.3) | 5467.9 (49.9) | 6176.3 (17.8) | 41.6 (288.7) | 218.8 (38.5) | 215.0 (163.5) | 225.6 (88.7) | 516.5 (74.3)

24. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time (AUC0-t) After First Dose of MSC2156119J: Regimen 2
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the LLQ. AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 3 | 4 | 6 | 7
h*ng/mL | 1771.5 (43.1) | 3665.3 (41.9) | 3794.2 (32.1) | 4659.6 (44.9) | 10818.0 (48.9) | 206.9 (92.6) | 310.5 (27.6) | 745.3 (130.8) | 1323.5 (57.3)

25. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time (AUC0-t) After First Dose of MSC2156119J: Regimen 3
Description: as for outcome 24
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- MSC2156119J 500 mg Fasted: Subjects were administered with micronized MSC2156119J 500 mg (capsule formulation) in the fasted state.
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 19 | 3 | 7 | 1 | 6 | 22
h*ng/mL | 4209.3 (33.4) | 3190.8 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 5667.3 (76.1) | 4980.9 (86.3) | 10355.6 (59.6) | 13352.6 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 15542.0 (41.9) | 7661.8 (66.7)

26. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Multiple Dose of MSC2156119J : Regimen 1
Description: as for outcome 24
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3
h*ng/mL | 7532.7 (19.1) | 14113.2 (32.1) | 18334.0 (19.4) | 18409.6 (14.3) | 56102.4 (73.7) | 82253.4 (10.1) | 44598.2 (80.7) | 2008.0 (344.0) | 4483.4 (284.9) | 3555.4 (116.3) | 4234.1 (40.3) | 13872.2 (62.3)

27. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Multiple Dose of MSC2156119J : Regimen 2
Description: as for outcome 24
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3 | 3 | 3 | 6 | 6
h*ng/mL | 4079.6 (71.1) | 5079.7 (116.0) | 4962.0 (33.3) | 7963.8 (34.0) | 36701.1 (26.1) | 375.2 (278.2) | 2056.6 (31.4) | 2562.0 (78.9) | 2899.0 (132.4)

28. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Multiple Dose of MSC2156119J : Regimen 3
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the LLQ. AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. Reporting group "MSC2156119J 1200 mg: Fasted" is not applicable for Multiple Dosing because only one subject was erroneously dosed with 1200 mg in fasted state as a single dose in Regimen 3. For multiple dose PK profile (Study Day 14), this subject was included in reporting group "MSC2156119J 1400 mg: Fed".
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- MSC2156119J 300 mg Fed: Subjects were administered with micronized MSC2156119J 300 mg (capsule formulation) with food.
Arm/Group | MSC2156119J 300 mg Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 17 | 3 | 6 | 4 | 18
h*ng/mL | 15694.9 (50.8) | 17498.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 20210.4 (33.5) | 17107.8 (3.2) | 27716.9 (58.6) | 39730.6 (29.5) | 18915.7 (87.5)

29. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) After Single Dose Of MSC2156119J: Regimen 1
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of AUC0-inf.
Groups:
- MSC2156119J 145 mg Fed: Subjects were administered with micronized MSC2156119J 145 mg (capsule formulation) with food.
- MSC2156119J 215 mg Fed: Subjects were administered with micronized MSC2156119J 215 mg with food.
- MSC2156119J 400 mg Fed: Subjects were administered with micronized MSC2156119J 400 mg (capsule formulation) with food.
- MSC2156119J 115 mg Fasted: Subjects were administered with non-micronized MSC2156119J 115 mg (capsule formulation) in the fasted state.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg Fed | MSC2156119J 215 mg Fed | MSC2156119J 300 mg Fed | MSC2156119J 400 mg Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) After Single Dose Of MSC2156119J: Regimen 2
Description: as for outcome 29
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 29
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) After Single Dose Of MSC2156119J: Regimen 3
Description: as for outcome 29
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 29
Arm/Group | MSC2156119J 300 mg Fed | MSC2156119J 500 mg Fasted | MSC2156119J 500 mg Fed | MSC2156119J 700 mg Fed | MSC2156119J 1000 mg Fed | MSC2156119J 1200 mg Fasted | MSC2156119J 1400 mg Fed | MSC2156119J 500 mg Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Single Dose of MSC2156119: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 5 | 6 | 3
h*ng/mL | 848.7 (24.3) | 1283.0 (23.9) | 1731.3 (14.9) | 2454.5 (15.4) | 3090.2 (61.2) | 5462.8 (49.9) | 6176.3 (17.8) | 94.0 (66.2) | 218.8 (38.5) | 259.3 (170.5) | 220.6 (93.4) | 515.3 (74.4)

33. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Single Dose of MSC2156119: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24, 48 hours post-dose on Day 1 Cycle 1
Population: PK analysis set included all subjects who had received at least 1 dose of MSC2156119J and who had provided at least 1 concentration of MSC2156119J measurement after the first dose. Here, "Number Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 3 | 3 | 4 | 7
h*ng/mL | 1771.5 (43.1) | 3657.3 (42.0) | 3794.2 (32.1) | 4659.6 (44.9) | 10786.4 (49.4) | 206.9 (92.6) | 306.1 (33.9) | 626.0 (96.5) | 1317.0 (58.3)

34. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Single Dose of MSC2156119: Regimen 3
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 18 | 2 | 6 | 1 | 6 | 22
h*ng/mL | 4206.5 (33.5) | NA (NA) — Data were not reported to reduce misunderstanding as 1 subject in "MSC2156119J 500 mg: Fasted arm" either took a wrong dose or intake was performed with a wrong mode of administration. | 5917.9 (74.8) | 7575.8 (24.6) | 11796.4 (48.1) | NA (NA) — Data were not reported to reduce misunderstanding as 1 subject in "MSC2156119J 1200 mg: Fasted arm" either took a wrong dose or intake was performed with a wrong mode of administration. | 15542.0 (41.9) | 7637.3 (66.7)

35. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Multiple Dose of MSC2156119: Regimen 1
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3
h*ng/mL | 2266.7 (29.5) | 4443.1 (28.1) | 5499.6 (7.0) | 8099.6 (18.0) | 13938.4 (50.9) | 18276.5 (12.4) | 12256.8 (49.1) | 585.3 (158.4) | 1241.2 (132.2) | 1011.1 (110.3) | 1434.2 (14.3) | 4658.2 (52.4)

36. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Multiple Dose of MSC2156119: Regimen 2
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24, 48 hours post-dose on Day 19 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 5 | 4 | 5 | 1 | 3 | 2 | 3 | 5 | 4
h*ng/mL | 3031.7 (55.8) | 7565.6 (35.0) | 5305.5 (62.6) | 9051.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 27760.2 (25.1) | 273.7 (909.0) | 2054.1 (33.3) | 1634.4 (103.5) | 3538.9 (64.9)

37. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve Within One Dosing Interval (AUCtau) After Multiple Dose of MSC2156119: Regimen 3
Description: as for outcome 10
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 3 | 1 | 17 | 3 | 6 | 4 | 13
h*ng/mL | 15597.6 (50.0) | 17498.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 20169.3 (33.5) | 21972.2 (42.9) | 27214.4 (59.4) | 39283.7 (28.0) | 27437.7 (51.7)

38. Secondary Outcome: Apparent Body Clearance (CL/f) After First Dose of MSC2156119J: Regimen 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from plasma, CL= Dose/AUC0-inf.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of CL/f.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Apparent Body Clearance (CL/f) After First Dose of MSC2156119J: Regimen 2
Description: as for outcome 38
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 38
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Apparent Body Clearance (CL/f) After First Dose of MSC2156119J: Regimen 3
Description: as for outcome 38
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 38
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After First Dose of MSC2156119J: Regimen 1
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by λz.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of Vz/f.
Groups:
- MSC2156119J 60 mg Fasted: Subjects were administered with non-micronized MSC2156119J 60 mg (capsule formulation) in the fasted state.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After First Dose of MSC2156119J: Regimen 2
Description: as for outcome 41
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 41
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After First Dose of MSC2156119J: Regimen 3
Description: as for outcome 41
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 41
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After Multiple Dose of MSC2156119J: Regimen 1
Description: as for outcome 41
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 41
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After Multiple Dose of MSC2156119J: Regimen 2
Description: as for outcome 41
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 41
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Secondary Outcome: Apparent Volume of Distribution (Vz/f) After Multiple Dose of MSC2156119J: Regimen 3
Description: as for outcome 41
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 41
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Single Dose of MSC2156119J: Regimen 1
Description: Apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant.
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Single Dose of MSC2156119J: Regimen 2
Description: as for outcome 47
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 47
Groups:
- MSC2156119J 115 mg Fed: Subjects were administered with non-micronized MSC2156119J 115 mg (capsule formulation) with food.
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Single Dose of MSC2156119J: Regimen 3
Description: as for outcome 47
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 47
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1200 mg: Fasted | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Multiple Dose of MSC2156119J: Regimen 1
Description: as for outcome 47
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 47
Arm/Group | MSC2156119J 30 mg: Fed | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 145 mg: Fed | MSC2156119J 215 mg: Fed | MSC2156119J 300 mg: Fed | MSC2156119J 400 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed | MSC2156119J 230 mg: Fasted
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Multiple Dose of MSC2156119J: Regimen 2
Description: as for outcome 47
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 19 Cycle 1
Population: as for outcome 47
Arm/Group | MSC2156119J 60 mg: Fed | MSC2156119J 100 mg: Fed | MSC2156119J 130 mg: Fed | MSC2156119J 175 mg: Fed | MSC2156119J 315 mg: Fed | MSC2156119J 30 mg: Fasted | MSC2156119J 60 mg: Fasted | MSC2156119J 115 mg: Fasted | MSC2156119J 115 mg: Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

52. Secondary Outcome: Apparent Terminal Rate Constant (λz) After Multiple Dose of MSC2156119J: Regimen 3
Description: as for outcome 47
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 47
Arm/Group | MSC2156119J 300 mg: Fed | MSC2156119J 500 mg: Fasted | MSC2156119J 500 mg: Fed | MSC2156119J 700 mg: Fed | MSC2156119J 1000 mg: Fed | MSC2156119J 1400 mg: Fed | MSC2156119J 500 mg: Fed (Tablet)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Absolute Change From Baseline in Cytoplasm and Membrane H-Score at Day 1 Cycle 2
Description: Histo score (H-score) is a composite score that comprises of intensity and percentage of staining and is used for assessing the amount of protein or phospho-protein present in a biopsy sample. The composite score obtained by H-score is derived by summing the percentages of cell staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+; where 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). The composite H-score ranges from 0 to 300, with a score of 0 representing the absence of any of the target protein and an H-score of 300 representing maximum staining and intensity of the target protein.
Time Frame: Baseline, Day 1 Cycle 2
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment. Here, "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 17 | 21 | 32
units on a scale
  Cytoplasm H-Score | -12.94 (84.614) | -31.43 (92.967) | 5.00 (72.513)
  Membrane H-Score | 3.53 (123.184) | 28.10 (75.407) | -10.00 (75.818)

54. Secondary Outcome: Fold Change From Baseline in Cytoplasm and Membrane H-Score at Day 1 Cycle 2
Description: Histo score (H-score) is a composite score that comprises of intensity and percentage of staining and is used for assessing the amount of protein or phospho-protein present in a biopsy sample. The composite score obtained by H-score is derived by summing the percentages of cell staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+; where 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). The composite H-score ranges from 0 to 300, with a score of 0 representing the absence of any of the target protein and an H-score of 300 representing maximum staining and intensity of the target protein. Fold change = on-treatment value/ baseline value
Time Frame: Baseline, Day 1 Cycle 2
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment. Here "Number of Participants analyzed" signifies those subjects who were evaluable for this outcome and "n" signifies those subjects who were evaluable in the specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 16 | 17 | 30
fold change
  Cytoplasm H-Score (n=16, 17, 30) | 1.05 (0.577) | 1.09 (0.570) | 1.12 (0.551)
  Membrane H-Score (n= 0, 4, 5) | NA (NA) — Fold change could not be calculated as there were no subjects with H-score baseline value of greater than 0. | 1.29 (0.934) | 1.23 (0.541)

55. Secondary Outcome: Number of Subjects With Monovalent Antagonist Antibody to Receptor MET (MetMAb) Score (MMS)
Description: MetMAb score was used to assess the tumor c-Met expression and ranged from 0 to 3, where a score of 0 corresponds to the lowest c-Met expression and a score of 3 corresponds to the highest c-Met expression in tumor tissue by immunohistochemistry.
Time Frame: Day 1 Cycle 2
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 42 | 45 | 62
subjects
  MMS Score 0 | 3 | 5 | 1
  MMS Score 1 | 9 | 7 | 12
  MMS Score 2 | 4 | 10 | 14
  MMS Score 3 | 2 | 2 | 8
  MMS Score Missing | 24 | 21 | 27

56. Secondary Outcome: Relative Percentage Change In Sum of Longest Diameter (SOLD) of Target Lesions to Post-Baseline Nadir
Description: The post-baseline nadir was defined as the the smallest SOLD recorded after baseline. The relative change (%) was derived based on the SOLD of target lesions as follows: 100* (SOLD at post-baseline nadir - baseline SOLD) / baseline SOLD.
Time Frame: Baseline, On Treatment (up to 153.3 weeks)
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment. Here "Number of Participants Analyzed" signifies those subjects who presented a measurable tumor at baseline and at least one post-baseline tumor assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 35 | 36 | 52
percent change | 25.67 (28.738) | 16.19 (22.055) | 18.87 (39.464)

57. Secondary Outcome: Number of Subjects With Best Overall Response (BOR)
Description: Number of subjects with BOR in each category (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) was reported. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: defined as at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD:defined as at least a 20% increase in sum of longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameter while on study.
Time Frame: Baseline up to 153.3 weeks
Population: Safety set included all subjects who had received at least 1 dose of MSC2156119J treatment.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 42 | 45 | 62
subjects
  CR | 0 | 0 | 0
  PR | 0 | 0 | 2
  SD | 12 | 10 | 12
  PD | 25 | 27 | 38
  Not evaluable | 5 | 8 | 10

58. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time (in months) between the first dosing day and radiographic PD or clinical PD (as recorded on the study termination form) or death, if death occurred within 12 weeks (84 days) after the last tumor assessment without documented progressive disease, whichever occurred first. Any subject with neither assessment of tumor progression, nor death within 12 weeks after last tumor assessment date was censored on the date of last tumor assessment.
Time Frame: Baseline up to 153.3 weeks
Population: as for outcome 53
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Number analyzed (Participants) | 41 | 45 | 62
months | 1.4 [1.3 to 1.4] | 1.3 [1.2 to 1.3] | 1.4 [1.3 to 1.4]

ADVERSE EVENTS:
Time Frame: Baseline up to 158.01 weeks
Arm/Group | MSC2156119J Regimen 1 | MSC2156119J Regimen 2 | MSC2156119J Regimen 3
Serious Adverse Events (participants affected / at risk) | 14/42 | 17/45 | 22/62
Other Adverse Events (participants affected / at risk) | 41/42 | 45/45 | 59/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC2156119J Regimen 1 (N=42) | MSC2156119J Regimen 2 (N=45) | MSC2156119J Regimen 3 (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 1 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 4
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 4
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 4 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 4
VOMITING (Gastrointestinal disorders) | 0 | 2 | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0
FAECALOMA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 0 | 1
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 1 | 0
DEVICE OCCLUSION (General disorders) | 1 | 0 | 0
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 1
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 0 | 1 | 0
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 2 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 1
ABDOMINAL WALL INFECTION (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
GANGRENE (Infections and infestations) | 1 | 0 | 0
KIDNEY INFECTION (Infections and infestations) | 1 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 1 | 0
WAIST CIRCUMFERENCE INCREASED (Investigations) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 2 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 1
VAGUS NERVE DISORDER (Nervous system disorders) | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 3
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 2 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC2156119J Regimen 1 (N=42) | MSC2156119J Regimen 2 (N=45) | MSC2156119J Regimen 3 (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 4 | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 5 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 2 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 1
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 0 | 0 | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 2 | 2 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 1
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0
DEAFNESS (Ear and labyrinth disorders) | 1 | 0 | 1
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 0 | 0
EAR SWELLING (Ear and labyrinth disorders) | 1 | 0 | 0
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 2 | 1 | 1
BASEDOW'S DISEASE (Endocrine disorders) | 0 | 1 | 0
THYROID DISORDER (Endocrine disorders) | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 2 | 0 | 4
DRY EYE (Eye disorders) | 0 | 0 | 2
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 1
BLEPHAROSPASM (Eye disorders) | 1 | 0 | 0
RETINAL PIGMENT EPITHELIOPATHY (Eye disorders) | 1 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 1 | 0
VITREOUS FLOATERS (Eye disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 12 | 10 | 16
NAUSEA (Gastrointestinal disorders) | 11 | 10 | 11
VOMITING (Gastrointestinal disorders) | 11 | 8 | 10
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 7 | 9
DIARRHOEA (Gastrointestinal disorders) | 7 | 6 | 6
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 5 | 6
ASCITES (Gastrointestinal disorders) | 1 | 6 | 6
DRY MOUTH (Gastrointestinal disorders) | 2 | 2 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 | 2
DYSPHAGIA (Gastrointestinal disorders) | 1 | 1 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 1 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1
MELAENA (Gastrointestinal disorders) | 2 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 2 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 1 | 0
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 1 | 0 | 0
ERUCTATION (Gastrointestinal disorders) | 1 | 0 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL SOUNDS ABNORMAL (Gastrointestinal disorders) | 1 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0 | 0
LIP SWELLING (Gastrointestinal disorders) | 0 | 1 | 0
NEUROGENIC BOWEL (Gastrointestinal disorders) | 1 | 0 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
RETCHING (Gastrointestinal disorders) | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 12 | 17 | 20
OEDEMA PERIPHERAL (General disorders) | 6 | 9 | 24
PYREXIA (General disorders) | 5 | 1 | 6
CHILLS (General disorders) | 2 | 1 | 4
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 4 | 1
MALAISE (General disorders) | 0 | 3 | 1
PERIPHERAL SWELLING (General disorders) | 3 | 0 | 1
ASTHENIA (General disorders) | 1 | 1 | 1
AXILLARY PAIN (General disorders) | 1 | 0 | 1
EARLY SATIETY (General disorders) | 0 | 0 | 2
GAIT DISTURBANCE (General disorders) | 0 | 0 | 2
LOCAL SWELLING (General disorders) | 1 | 1 | 0
OEDEMA (General disorders) | 0 | 1 | 1
PAIN (General disorders) | 0 | 0 | 2
CATHETER SITE ERYTHEMA (General disorders) | 1 | 0 | 0
FEELING COLD (General disorders) | 0 | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 0 | 1
LOCALISED OEDEMA (General disorders) | 0 | 0 | 1
SENSATION OF FOREIGN BODY (General disorders) | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 5 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 0 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 3 | 7
ORAL CANDIDIASIS (Infections and infestations) | 1 | 4 | 2
PNEUMONIA (Infections and infestations) | 0 | 1 | 3
SINUSITIS (Infections and infestations) | 1 | 2 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1 | 0
EAR INFECTION (Infections and infestations) | 1 | 0 | 0
HORDEOLUM (Infections and infestations) | 0 | 0 | 1
INFECTED FISTULA (Infections and infestations) | 1 | 0 | 0
NAIL BED INFECTION FUNGAL (Infections and infestations) | 1 | 0 | 0
ONYCHOMYCOSIS (Infections and infestations) | 1 | 0 | 0
PAROTITIS (Infections and infestations) | 0 | 0 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 1
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1
UROSEPSIS (Infections and infestations) | 0 | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 3 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 | 0 | 1
FEEDING TUBE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
NAIL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
STOMA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 | 5 | 8
LIPASE INCREASED (Investigations) | 3 | 4 | 2
TRANSAMINASES INCREASED (Investigations) | 1 | 1 | 7
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1 | 6
BLOOD CREATININE INCREASED (Investigations) | 3 | 0 | 5
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 3 | 2
BREATH SOUNDS ABNORMAL (Investigations) | 2 | 1 | 3
WEIGHT DECREASED (Investigations) | 0 | 1 | 3
AMYLASE INCREASED (Investigations) | 2 | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 2
HAEMOGLOBIN INCREASED (Investigations) | 0 | 2 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 2 | 0
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 0 | 0 | 2
WEIGHT INCREASED (Investigations) | 1 | 1 | 0
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 1 | 0 | 0
BLOOD CREATINE INCREASED (Investigations) | 0 | 0 | 1
BLOOD GLUCOSE DECREASED (Investigations) | 1 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0 | 0
BLOOD PRESSURE DIASTOLIC ABNORMAL (Investigations) | 0 | 0 | 1
BLOOD UREA INCREASED (Investigations) | 0 | 1 | 0
ELECTROCARDIOGRAM PR SHORTENED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 1
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 0 | 0 | 1
HAEMATOCRIT INCREASED (Investigations) | 0 | 1 | 0
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 1 | 0
PEDAL PULSE ABNORMAL (Investigations) | 0 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 1 | 0
WAIST CIRCUMFERENCE INCREASED (Investigations) | 0 | 0 | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 | 5 | 27
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 8 | 6 | 11
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 4 | 9
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 2 | 8
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 | 3 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 5 | 4
HYPOKALAEMIA (Investigations) | 3 | 3 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 3
CACHEXIA (Metabolism and nutrition disorders) | 1 | 1 | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 2
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
JOINT ANKYLOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
TUMOUR INVASION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 3 | 5 | 7
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 4 | 4
HEADACHE (Nervous system disorders) | 1 | 2 | 4
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 2 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 3 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 3
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
TREMOR (Nervous system disorders) | 0 | 1 | 1
AKATHISIA (Nervous system disorders) | 0 | 0 | 1
BALANCE DISORDER (Nervous system disorders) | 0 | 1 | 0
DIZZINESS POSTURAL (Nervous system disorders) | 0 | 1 | 0
DYSKINESIA (Nervous system disorders) | 0 | 0 | 1
HYPOGEUSIA (Nervous system disorders) | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 1
NEURALGIA (Nervous system disorders) | 0 | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 1
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 4 | 1 | 6
ANXIETY (Psychiatric disorders) | 1 | 0 | 3
AGITATION (Psychiatric disorders) | 0 | 0 | 3
DELIRIUM (Psychiatric disorders) | 1 | 1 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0
EMOTIONAL DISTRESS (Psychiatric disorders) | 0 | 0 | 1
FLAT AFFECT (Psychiatric disorders) | 0 | 0 | 1
RESTLESSNESS (Psychiatric disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 1 | 4
PROTEINURIA (Renal and urinary disorders) | 1 | 2 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 2 | 0
DYSURIA (Renal and urinary disorders) | 2 | 1 | 0
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 1
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 0
NEUROGENIC BLADDER (Renal and urinary disorders) | 1 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 1
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 1
RENAL ATROPHY (Renal and urinary disorders) | 0 | 1 | 0
RENAL HYPERTROPHY (Renal and urinary disorders) | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 1
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 0 | 1
URINARY HESITATION (Renal and urinary disorders) | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
SCROTAL OEDEMA (Reproductive system and breast disorders) | 1 | 0 | 2
NIPPLE PAIN (Reproductive system and breast disorders) | 0 | 2 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 1
BREAST MASS (Reproductive system and breast disorders) | 0 | 0 | 1
BREAST SWELLING (Reproductive system and breast disorders) | 1 | 0 | 0
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 | 0 | 1
DYSPAREUNIA (Reproductive system and breast disorders) | 0 | 0 | 1
NIPPLE DISORDER (Reproductive system and breast disorders) | 0 | 1 | 0
PENILE OEDEMA (Reproductive system and breast disorders) | 0 | 0 | 1
SCROTAL SWELLING (Reproductive system and breast disorders) | 0 | 1 | 0
TESTICULAR SWELLING (Reproductive system and breast disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 12
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 3 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 3
HYPOTENSION (Vascular disorders) | 1 | 0 | 2
HYPERTENSION (Vascular disorders) | 1 | 1 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 1
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
It was not possible to calculate data for PK parameters such as t1/2, AUC0-inf, CL/f, Vz/f, λz because dosing interval was too small compared to the long half-life to characterize terminal phase rate constant, which is needed for the calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No